CLINICAL TRIAL: NCT01343511
Title: Phase Ι/Π Study of Stem Cell Therapy in Patients With Autism
Brief Title: Safety and Efficacy of Stem Cell Therapy in Patients With Autism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Collaborators: Shandong Jiaotong Hospital (Unknown); Association for the Handicapped Of Jinan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BKCR-AUTISM-1.0(2009)
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Autism
Keywords: Autism; human cord blood mononuclear cells; human umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation plus hCB-MNCs treatment (Experimental): Participants will be given rehabilitation therapy plus human cord blood mononuclear cells transplantation with a 6 months follow-up.
  Interventions: Biological: human cord blood mononuclear cells
- Rehabilitation plus hCB-MNCs and hUC-MSCs therapy (Experimental): Participants will be given rehabilitation therapy plus combination of hCB-MNCs together with hUC-MSCs transplantation with a 6 months follow-up.
  Interventions: Biological: human cord blood mononuclear cells and human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: human cord blood mononuclear cells — Participants will be given rehabilitation therapy plus hCB-MNCs transplantation.
  Other Names: Group 1
  Arms: Rehabilitation plus hCB-MNCs treatment
Biological: human cord blood mononuclear cells and human umbilical cord mesenchymal stem cells — Participants will be given rehabilitation therapy plus and hCB-MNCs and hUC-MSCs transplantation.
  Other Names: Group 2
  Arms: Rehabilitation plus hCB-MNCs and hUC-MSCs therapy

SUMMARY:
Autism is one of those disorders in Autism spectrum disorders (ASD), which characterized by social interaction abnormalities, impaired verbal and non-verbal communication, and repetitive, obsessive behavior, while the therapeutic effect of current treatments remains limited progress .Neural hypoperfusion and immune deregulation are the two key pathologies associated with Autism. Human umbilical cord mesenchymal stem cells (hUC-MSCs) and human cord blood mononuclear cells (hCB-MNCs) have been shown to have the ability to modulate the immune response and enhance angiogenesis, suggesting the novel and promising therapeutic strategy. In this study, the safety and efficacy of hUC-MSCs and hCB-MNCs transplantation will be evaluated in patients with Autism.

DETAILED DESCRIPTION:
To investigate the safety and efficacy of human cord blood mononuclear cells and human umbilical cord mesenchymal stem cells transplantation in patients of Autism.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3 and 12 years.
* DSM-IV diagnosis of Autistic Disorder.
* Total score of CARS ≥ 30.
* Parents or legal guardian willing to sign the ICF.

Exclusion Criteria:

* Any history of hypersensitivity to serum products, or other known drug and food allergy.
* History of prior or current DSM-IV psychotic disorder (e.g., schizophrenia, bipolar disorder, other psychosis), Pervasive Developmental Disorder not otherwise specified (PDD NOS), Asperger's, or Rett's.
* History of Epileptic seizure activity in the past 6 months.
* Autism caused by seizure disorders (active), cerebrovascular disease or brain trauma.
* The global autism ratings are assessed as being absent, minimal or mild.
* Existing moderate or severe extrapyramidal symptoms (EPS) or history of tardive dyskinesia.
* Subjects who have displayed significant self-injurious behavior (children who have caused visible harm to themselves).
* HIV+
* Acute and chronic hepatitis.
* Autoimmune disease, e.g. lupus erythematosus, multiple sclerosis.
* Severe pulmonary and hematological disease, malignancy or hypo-immunity.
* Currently undertaking other treatment that may affect the safety/efficacy of stem cells.
* Enrollment in other trials in the last 3 months.
* Other criteria the investigator consider improper for inclusion.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale，CARS | 6 months after treatment
Clinical Global Impression Scale，CGI | 6 months after treatment

SECONDARY OUTCOMES:
Aberrant Behavior Checklist，ABC | 6 months after treatment
Adverse Event and Serious Adverse Event | 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Lv, Principal Investigator — Shandong Jiaotong Hospital
Locations (1):
- Shandong Jiaotong Hospital, Jinan, Shandong, China

REFERENCES:
- [Result] Liu M, Sun LW, LV YT, Huan Y, Ge RC, Cao YL, Guo CQ, Chen XW. Stem cells for treatment of autism: Safety and efficacy. Zhongguo Zuzhi Gongcheng Yanjiu yu Linchuang Kangfu. 2010;14(32): 5967-5970.
- [Derived] Lv YT, Zhang Y, Liu M, Qiuwaxi JN, Ashwood P, Cho SC, Huan Y, Ge RC, Chen XW, Wang ZJ, Kim BJ, Hu X. Transplantation of human cord blood mononuclear cells and umbilical cord-derived mesenchymal stem cells in autism. J Transl Med. 2013 Aug 27;11:196. doi: 10.1186/1479-5876-11-196. PMID 23978163